CLINICAL TRIAL: NCT07335081
Title: A Randomized, Multicenter, Open-label Clinical Study Using Peripheral Blood Circulating Tumor DNA to Evaluate the Efficacy of Preoperative Treatment With Pyrotinib + Trastuzumab + Docetaxel Versus Pertuzumab + Trastuzumab + Docetaxel in Early or Locally Advanced HER2-positive Breast Cancer
Brief Title: ctDNA in HER2+ EBC Neoadjuvant Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC2401
Record Dates: First submitted 2025-12-21; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant therapy; HER2 positive; ctDNA
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; pertuzumab; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrotinib-initiated arm (Experimental): two cycles of docetaxel + trastuzumab + pyrotinib followed by two cycles of docetaxel + trastuzumab + pertuzumab
  Interventions: Drug: pyrotinib; Drug: pertuzumab; Drug: trastuzumab; Drug: docetaxel
- Pertuzumab-initiated arm (Active Comparator): four cycles of docetaxel + trastuzumab + pertuzumab
  Interventions: Drug: pertuzumab; Drug: trastuzumab; Drug: docetaxel

INTERVENTIONS:
Drug: pyrotinib — pyrotinib 320mg p.o. qd
  Arms: Pyrotinib-initiated arm
Drug: pertuzumab — pertuzumab ivgtt q3w, 840mg for initiation, 420mg for maintenance
Drug: trastuzumab — trastuzumab ivgtt q3w, 8mg/kg for initiation, 6mg/kg for maintenance
Drug: docetaxel — docetaxel ivgtt q3w, 80-100mg/m2

SUMMARY:
This study is a randomized, open-label, multicenter clinical study for patients with early or locally advanced (T≥2cm, N0-3, M0) HER2-positive breast cancer, aiming to compare the peripheral blood ctDNA clearance of neoadjuvant pyrotinib + trastuzumab + docetaxel and pertuzumab + trastuzumab + docetaxel for one course and to evaluate the therapeutic effectiveness of four courses of neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed with Stage II-III HER2+ breast cancer (primary diameter >2cm)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Intact renal, hepatic, bone marrow and cardiac functions including baseline left ventricular ejection fraction (LVEF) ≥ 55% measured by echocardiography
* No prior treatment

Exclusion Criteria:

* Bilateral or metastatic breast cancer
* History of other malignancies
* Severe cardiovascular disease
* Allergic to any of the regimens

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance after one cycle neoadjuvant treatment | 3 months after neoadjuvant treatment initation
  The rate of ctDNA clearance after first cycle of neoadjuvant treatment

SECONDARY OUTCOMES:
ctDNA clearance after two cycle neoadjuvant treatment | 3 months after neoadjuvant treatment initation
  The rate of ctDNA clearance after first two cycles of neoadjuvant treatments
pCR rate | 6 months after neoadjuvant treatment initation
  After completion of neoadjuvant therapy and surgery, no residual invasive carcinoma in the evaluation of hematoxylin and eosin stained mamtectomy samples and all ipsilateral lymph node samples
bpCR rate | 6 months after neoadjuvant treatment initation
  After completion of neoadjuvant therapy and surgery, no residual invasive carcinoma in the evaluation of hematoxylin and eosin stained breast samples
ORR | 6 months after neoadjuvant treatment initation
  The proportion of patients whose tumor volume shrinks to a prespecified value and is able to maintain the minimum time limit, defined as the sum of the proportion of complete response (CR) and partial response (PR, with a reduction in tumor length and diameter greater than 30%).
EFS | 2 years after surgery
  The time interval from randomization to the first recording of the following events: disease progression (before surgery), as determined by investigator reference RECIST1.1, combined with clinical evaluation, final judgment; postoperative disease recurrence (local, regional, distal, or contralateral); second primary malignancy; Death from any cause
DFS | 2 years after surgery
  The time interval from the first date of disease-free (i.e., the date of surgery) to the first recording of the following events; Postoperative disease recurrence (local, regional, distal, or contralateral); second primary malignancy; Death from any cause.
OS | 5 years after surgery
  Time interval from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China